CLINICAL TRIAL: NCT07238855
Title: Effect of Isometric Hand Grip Exercises Using a Dynamometer on Arteriovenous Fistula Maturation and Patency in Hemodialysis Patients
Brief Title: Effect of Isometric Hand Grip Exercises Using a Dynamometer on AV Fistula Maturation and Patency in Hemodialysis Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Mona Zidan, Resident of Internal Medicine and Nephrology, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MS.23.01.2266
Record Dates: First submitted 2025-11-16; First posted 2025-11-20 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Chronic Kidney Failure; End-Stage Renal Disease; Arteriovenous Fistula
Keywords: Arteriovenous fistula maturation; Arteriovenous fistula patency; Hemodialysis vascular access; Chronic kidney disease; End-stage renal disease; Hand-grip exercise; Isometric muscle exercise; Dynamometer training
MeSH Terms: conditions — Kidney Failure, Chronic; Arteriovenous Fistula; Renal Insufficiency, Chronic

STUDY DESIGN:
Intervention Model Description: Two-arm parallel randomized controlled study comparing standard postoperative care versus a structured isometric hand-grip exercise program using a dynamometer in adult hemodialysis patients with a surgically created arteriovenous fistula.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group - Standard Postoperative Care (No Intervention): Participants in this arm receive the standard postoperative care provided after the creation of an arteriovenous fistula for hemodialysis. They do not perform any structured exercise program. Routine follow-up assessments, including Doppler ultrasound evaluation of fistula diameter, blood flow, and blood flow velocity, are conducted at baseline and after six weeks.
- Hand-Grip Exercise Group - Isometric Training With Dynamometer (Experimental): Participants in this arm receive standard postoperative care plus a structured isometric hand-grip exercise program using a hand-held dynamometer. The intervention consists of adjusting the dynamometer grip to hand size, positioning the arm at a ninety-degree angle, and performing three maximal-effort squeezes repeated to calculate average grip strength. Exercises are performed regularly for six weeks. Doppler ultrasound measurements of fistula diameter, vein caliber, blood flow, and blood flow velocity are obtained at baseline and after six weeks to evaluate maturation and patency.
  Interventions: Behavioral: Isometric Hand-Grip Exercise Training Using a Hand Dynamometer

INTERVENTIONS:
Behavioral: Isometric Hand-Grip Exercise Training Using a Hand Dynamometer — Participants perform a structured isometric hand-grip exercise program using a hand-held dynamometer for six weeks after creation of an arteriovenous fistula for hemodialysis. The grip handle is adjusted to the size of the hand, the elbow is flexed to a ninety-degree angle, and the participant performs repeated maximal voluntary hand-grip contractions according to a standardized schedule. Training is added to usual postoperative care and is monitored during follow-up visits.
  Arms: Hand-Grip Exercise Group - Isometric Training With Dynamometer

SUMMARY:
Patients with chronic kidney failure who require hemodialysis depend on a surgically created connection between an artery and a vein in the arm, known as an arteriovenous fistula. This connection allows blood to flow at a high enough rate for effective hemodialysis treatment. However, many arteriovenous fistulas do not enlarge or strengthen adequately after surgery, a process known as maturation. When maturation fails, the fistula may not provide enough blood flow, leading to delays in hemodialysis, repeated procedures, or the need for temporary catheters. Improving the maturation of arteriovenous fistulas is therefore essential for patient safety, comfort, and the long-term success of hemodialysis.

Isometric hand-grip exercises, such as repeatedly squeezing a hand-held dynamometer, may help increase blood flow to the arm and stimulate the blood vessels that are part of the fistula. These exercises require the muscles to contract without changing length, which can encourage enlargement of the vein and the development of new small blood vessels in the forearm. Previous research suggests that improving hand-grip strength may support better vein remodeling and improved blood flow, both of which are important for fistula maturation.

This study is designed to evaluate whether performing a structured program of isometric hand-grip exercises using a dynamometer can enhance the maturation and long-term openness (patency) of arteriovenous fistulas in adults receiving hemodialysis. Participants are randomly assigned to one of two groups: a control group that receives routine postoperative care, and an exercise group that performs hand-grip exercises for six weeks. All participants undergo ultrasound imaging of the fistula before starting the study and again after six weeks. The ultrasound measurements include fistula size, vein diameter, blood flow, and blood flow velocity.

The goal of this study is to determine whether a simple, low-cost exercise intervention can help arteriovenous fistulas mature more successfully and reduce the need for additional procedures.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 to 75 years
* End-stage renal disease requiring hemodialysis
* Patients undergoing hemodialysis through a surgically created arteriovenous fistula
* Ability to provide written informed consent

Exclusion Criteria:

* Failure or refusal to provide written informed consent
* Amputation of the arm or fingers
* Significant osteoarthritis of the hand or wrist
* Severe physical disability preventing exercise performance
* Active infection or ongoing hospitalization
* Known underlying malignancy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2023-02-15 (Actual); Primary Completion 2024-01-15 (Actual); Study Completion 2024-02-15 (Actual)

PRIMARY OUTCOMES:
Change in arteriovenous fistula blood flow volume measured by Doppler ultrasound | Baseline and six weeks after starting the hand-grip exercise program or standard care
  Blood flow volume through the arteriovenous fistula (milliliters per minute) will be measured using duplex Doppler ultrasound at the outflow vein. The primary metric is the change in blood flow volume from baseline (before starting the hand-grip exercise program or standard care) to six weeks. Change will be calculated as the value at six weeks minus the baseline value for each participant.

SECONDARY OUTCOMES:
Change in arteriovenous fistula vein diameter measured by Doppler ultrasound | Baseline and six weeks after starting the hand-grip exercise program or standard care
  Vein diameter of the arteriovenous fistula (millimeters) will be measured using duplex Doppler ultrasound at the inflow and outflow segments. The metric is the change in vein diameter from baseline to six weeks.
Change in hand-grip muscle strength of the dominant hand | Baseline and six weeks after starting the hand-grip exercise program or standard care
  Maximum isometric hand-grip strength (kilograms or newtons) will be assessed using a calibrated hand-held dynamometer. Each participant performs three maximal voluntary contractions with the dominant hand, and the mean of the three values is recorded. The metric is the change in hand-grip strength from baseline to six weeks.
Clinical usability of the arteriovenous fistula for hemodialysis | Assessed at six weeks after starting the hand-grip exercise program or standard care
  Proportion of participants whose arteriovenous fistula can be used successfully for routine hemodialysis, defined as achieving two-needle cannulation with the prescribed blood flow rate during at least three consecutive hemodialysis sessions without access failure or thrombosis.

CONTACTS AND LOCATIONS:
Locations (1):
- Mansoura Nephrology and Dialysis Unit - Mansoura University Hospitals, Al Mansurah, Dakahlia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No